CLINICAL TRIAL: NCT04731350
Title: Effect of Extra Corporeal Shock Wave Versus Dexamethasone Iontophoresis in Treatment of Knee Osteoarthritis
Brief Title: Shock Wave Versus Iontophoresis in Treatment of Subjects With Knee Osteoarthritis
Acronym: Shockwave
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shimaa Taha Abu El Kasem, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/012/002633
Record Dates: First submitted 2021-01-16; First posted 2021-01-29 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Iontophoresis; Exercise

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Shock wave(A) (Experimental): subjects will recive radial extracorporeal shock wave (2000 shock/session, 10Hz and EFD 0.178 mJ/mm²) on knee joints once per week for four weeks in addition to strengthening exercise
  Interventions: Device: radial extracorporeal shock wave; Other: Exercise
- Iontophoresis (B) (Experimental): subjects will recive dexamethasone iontophoresis on knee joints once per week for four weeks in addition to strengthening exercise
  Interventions: Device: iontophoresis; Other: Exercise
- Control (C) (Other): stregnthening exercise;straight leg raising exercisein which the patients were positioned in the crook lying position with the unexercised limb was the flexed one then the patients were asked to contract the quadriceps muscle and elevate the limb to 45º and hold for 6 seconds, slowly lower the limb and then relax for 6 seconds, three sets of 10 repetitions were don ,Isometric quadriceps contraction (quadriceps drill) in full knee extension maintained for 5 seconds, followed by a 5-second rest; the exercise was performed for 20 repetitions per session .treatment once per week for four weeks
  Interventions: Other: Exercise

INTERVENTIONS:
Device: radial extracorporeal shock wave — Radial shock wave device, Swiss DolorClast (EMS Electro Medical Systems, Nyon, Switzerland)
  Arms: Shock wave(A)
Device: iontophoresis — Iontophoretic drug delivery system (phoresors II auto model PM850 IOMED):
  Arms: Iontophoresis (B)
Other: Exercise — strengthening exercise

SUMMARY:
Both extra corporeal shock wave and dexamethasone iontophoresisare effective in treatment of knee osteoarthritis but which one is more effective is not clear yet . so the purpose of this study was to investigate and compare between the effect of shock wave and iontophoresis in treatment of knee osteoarthritis . it was hypothesized that there will be no difference between the effect of shock wave and iontophoresis on treatment of knee osteoarthritis.

DETAILED DESCRIPTION:
60 subjects with grade II knee osteoarthritis will be recruited from outpatient clinic of faculty of physical therapy and then they will be assigned randomly by sealed envelope into three groups ;group A (shock wave group) will received radial extracorporeal shock wave ,group B (Iontophoresis group ) will receive deaxamthasone iontophoresis and group c (control group) will receive traditional tratment ( stregnthening exerciseces) all treatment will be once session per week for four weeks .pain intensity ,knee ROM and knee injury and osteoarthritis outcome score physical function short (KOOS-PS).

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic knee OA for at least 3 months according to clinical criteria of American College of Rheumatology
2. Radiologic findings had to be compatible with knee OA, with kelgren and Lawrence (K-L) grade 2 in a simple X ray .
3. Tenderness on medial tibial plateau
4. Intensity of pain: visual analogue scale equal to 5 or greater
5. Failure of two or more types of previous conservative treatment (medication, anti-inflammatory drugs, physical therapy, stretching, acupuncture, orthotics and others)

Exclusion Criteria:

1. Neuorological and vestibular system disorder, systematic inflammatory disease, steroid injections in the last six months
2. Any contraindication to magnetic resonance imaging or radiography, or trauma history on knee
3. history of previous knee surgery -

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
visual analogue scale (VAS) | change from baseline to immediately pre treatment and from pre treatment to immediately post treatment
  pain intensity will be assessed by using visual analogue scale

SECONDARY OUTCOMES:
knee range of motion (ROM) | change from baseline to immediately pre treatment and from pre treatment to immediately post treatment
  electronic geniometer
knee injury and osteoarthritis outcome score physical function short (KOOS-PS) | change from baseline to immediately pre treatment and from pre treatment to immediately post treatment
  knee function by using KOOS-PS questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy ,Cairo University, Giza, Egypt